CLINICAL TRIAL: NCT01554852
Title: Randomised Comparisons, in Myeloma Patients of All Ages, of Thalidomide, Lenalidomide, Carfilzomib and Bortezomib Induction Combinations, and of Lenalidomide and Combination Lenalidomide Vorinostat as Maintenance (Myeloma XI)
Brief Title: Use of Thalidomide, Lenalidomide, Carfilzomib, Bortezomib and Vorinostat in the Initial Treatment of Newly Diagnosed Multiple Myeloma Patients
Acronym: Myeloma XI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leeds (Other)
Collaborators: Celgene (Industry); Merck Sharp & Dohme LLC (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number: 2009-010956-93
Record Dates: First submitted 2012-02-21; First posted 2012-03-15 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Multiple Myeloma
Keywords: myeloma; lenalidomide; Revlimid; cyclophosphamide; dexamethasone; bortezomib; Velcade; vorinostat; Zolinza; stem cell; carfilzomib; Kyprolis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Neoadjuvant Therapy; Cyclophosphamide; Lenalidomide; Dexamethasone; cone rod homeobox protein; Clinical Protocols; Thalidomide; carfilzomib; Bortezomib; Maintenance; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive pathway (Active Comparator): The intensive pathway is aimed at younger and fitter patients who will receive the standard dose of chemotherapy. The initial treatments will be followed by high-dose chemotherapy with a stem cell transplant which is generally standard practice.
  Participants receive one treatment from each following stage in intensive pathway, depending on what they are randomised to (Protocol v6.0):
  1. Induction treatment:
     1. CRD regimen - cyclophosphamide, lenalidomide, dexamethasone
     2. CTD regimen - cyclophosphamide, thalidomide, dexamethasone
     3. CCRD regimen - carfilzomib, cyclophosphamide, lenalidomide, dexamethasone
  2. Consolidation treatment (depending on response to induction treatment):
     1. VCD regimen - bortezomib, cyclosphosphamide, dexamethasone
     2. No consolidation treatment
  3. High-dose therapy and stem cell transplant
  4. Maintenance treatment:
     1. Lenalidomide maintenance
     2. No maintenance
     3. Lenalidomide plus vorinostat maintenance (Protocol v5.0 only)
  Interventions: Drug: Induction (intensive pathway) - cyclophosphamide, lenalidomide, & dexamethasone (CRD) regimen; Drug: Induction (intensive pathway) - cyclophosphamide, thalidomide, & dexamethasone (CTD) regimen; Drug: Induction (intensive pathway) - carfilzomib, cyclophosphamide, lenalidomide, & dexamethasone (CCRD) regimen; Drug: Consolidation (intensive & non-intensive pathways) - bortezomib, cyclophosphamide, & dexamethasone (VCD) regimen; Drug: Maintenance (intensive & non-intensive pathways) - lenalidomide maintenance; Drug: Maintenance (intensive & non-intensive pathways - protocol v5.0 only) - lenalidomide plus vorinostat maintenance; Drug: High dose melphalan therapy and autologous stem cell transplant (intensive pathway only)
- Non-intensive pathway (Active Comparator): The non-intensive pathway is aimed at participants who are not deemed suitable for the stem cell transplant, and will receive lower doses of some of the drugs.
  Interventions in each stage of non-intensive pathway (depending on what the participant has been randomised to) - from Protocol v6.0:
  1. Induction treatment
     1. CRDa regimen - cyclophosphamide, lenalidomide, dexamethasone attenuated
     2. CTDa regimen - cyclophosphamide, thalidomide, dexamethasone attenuated
  2. Consolidation treatment (depending on participant's response to induction treatment):
     1. VCD regimen - bortezomib, cyclosphosphamide, dexamethasone
     2. No consolidation treatment
  3. Maintenance treatment
     1. Lenalidomide maintenance
     2. No maintenance
     3. Lenalidomide plus vorinostat maintenance (*for participants recruited under Protocol v5.0 only*)
  Interventions: Drug: Induction (non-intensive pathway) - cyclophosphamide, lenalidomide, & dexamethasone attenuated (CRDa) regimen; Drug: Induction (non-intensive pathway) - cyclophosphamide, thalidomide, & dexamethasone attenuated (CTDa) regimen; Drug: Consolidation (intensive & non-intensive pathways) - bortezomib, cyclophosphamide, & dexamethasone (VCD) regimen; Drug: Maintenance (intensive & non-intensive pathways) - lenalidomide maintenance; Drug: Maintenance (intensive & non-intensive pathways - protocol v5.0 only) - lenalidomide plus vorinostat maintenance

INTERVENTIONS:
Drug: Induction (intensive pathway) - cyclophosphamide, lenalidomide, & dexamethasone (CRD) regimen — Days 1 & 8 - cyclophosphamide 500 mg PO Days 1-21 - lenalidomide 25 mg daily PO Days 1-4 & 12-15 - dexamethasone 40 mg daily PO This cycle is repeated every 28 days
  Other Names: Revlimid (lenalidomide)
  Arms: Intensive pathway
Drug: Induction (intensive pathway) - cyclophosphamide, thalidomide, & dexamethasone (CTD) regimen — Days 1,8,15 (i.e. weekly) - cyclophosphamide 500 mg PO Continuously - thalidomide 50 mg hard capsules. Initially 100 mg daily PO for 3 weeks, increasing to 200 mg daily PO Days 1-4 and 12-15 - dexamethasone 40 mg daily PO The cycle is repeated every 21 days
  Arms: Intensive pathway
Drug: Induction (intensive pathway) - carfilzomib, cyclophosphamide, lenalidomide, & dexamethasone (CCRD) regimen — Days 1 & 8 - cyclophosphamide 500 mg PO Days 1 & 2, 8 & 9, 15 & 16 - carfilzomib 20*/36 mg/m2** IV (*carfilzomib 20 mg/m2 is only administered on days 1 and 2 of cycle 1; **carfilzomib will be dose capped at a body surface area of 2.2 m2) Days 1-21 - lenalidomide 25 mg daily PO Days 1-4, 8, 9 & 15, 16 - dexamethasone 40 mg daily PO This cycle is repeated every 28 days
  Other Names: Kyprolis (carfilzomib); Revlimid (lenalidomide)
  Arms: Intensive pathway
Drug: Induction (non-intensive pathway) - cyclophosphamide, lenalidomide, & dexamethasone attenuated (CRDa) regimen — Days 1 & 8 - cyclophosphamide 500 mg PO Days 1-21 - lenalidomide 25 mg daily PO Days 1-4 & 15-18 - dexamethasone 20 mg daily PO This cycle is repeated every 28 days
  Other Names: Revlimid (lenalidomide)
  Arms: Non-intensive pathway
Drug: Induction (non-intensive pathway) - cyclophosphamide, thalidomide, & dexamethasone attenuated (CTDa) regimen — Days 1, 8, 15, 22 (weekly) - cyclophosphamide 500 mg PO Continuously - thalidomide 50 mg hard capsules; initially 50 mg daily PO for 4 weeks, increasing every 4 weeks by 50 mg increments to 200 mg daily PO Days 1-4 & 15-18 - dexamethasone 20 mg daily PO This cycle is repeated every 28 days
  Arms: Non-intensive pathway
Drug: Consolidation (intensive & non-intensive pathways) - bortezomib, cyclophosphamide, & dexamethasone (VCD) regimen — Days 1, 4, 8 & 11 - bortezomib 1.3 mg/m2 SC or IV Days 1, 8, 15 - cyclophosphamide 500 mg PO Days 1-2, 4-5, 8-9 & 11-12 - dexamethasone 20 mg daily PO This cycle is repeated every 21 days
  Other Names: Velcade (bortezomib)
Drug: Maintenance (intensive & non-intensive pathways) - lenalidomide maintenance — Days 1-21 - lenalidomide 10 mg daily PO This cycle is repeated every 28 days
  Other Names: Revlimid (lenalidomide)
Drug: Maintenance (intensive & non-intensive pathways - protocol v5.0 only) - lenalidomide plus vorinostat maintenance — Days 1-21 - lenalidomide 10 mg daily PO Days 1-7 & 15-21 - vorinostat 300mg PO This cycle is repeated every 28 days
  Other Names: Revlimid (lenalidomide); Zolinza (vorinostat)
Drug: High dose melphalan therapy and autologous stem cell transplant (intensive pathway only) — High dose melphalan therapy and autologous stem cell transplant to be given as per local practice
  Arms: Intensive pathway

SUMMARY:
The purpose of this study is to compare a standard chemotherapy regimen of cyclophosphamide, dexamethasone plus thalidomide with a newer regimen of cyclophosphamide, dexamethasone plus lenalidomide with or without carfilzomib.

Patients who do not have the best response to their initial treatment may then also be given a combination of cyclophosphamide, dexamethasone plus bortezomib.

Patients who are relatively fit may, on their doctor's advice, go on to receive more intensive chemotherapy, supported with a transplant of their own blood cells. This is standard treatment which patients may be offered anyway even if they didn't take part in this study.

After maximal response has been achieved with the treatment described above, and as long as the myeloma has not got worse, patients will be treated with either long-term lenalidomide, lenalidomide with vorinostat, or receive no further treatment, with close observation.

DETAILED DESCRIPTION:
The last ten years has seen the introduction of a number of effective new anti-myeloma agents into the clinical arena. These agents have been shown to be highly effective in the relapse setting and now are being introduced as treatment earlier in the disease course.

This study aims to address in the randomised setting some of the key questions concerning the use of thalidomide, bortezomib, lenalidomide, carfilzomib and vorinostat in the initial treatment of multiple myeloma patients.

Newly diagnosed patients of all ages with symptomatic myeloma requiring treatment are eligible.

For initial treatment, thalidomide in combination with cyclophosphamide and dexamethasone, the UK gold standard, will be compared with the newer combination of lenalidomide, cyclophosphamide and dexamethasone with or without carfilzomib.

For patients with a sub-optimal response to initial therapy, the response to the proteasome inhibitor bortezomib will be assessed, as previous studies have demonstrated that it is able to induce responses and improve progression-free and overall survival in patients resistant to standard chemotherapy. Patients young and fit enough to tolerate an autologous transplant will then proceed to high dose melphalan with peripheral blood stem cell rescue and then on to maintenance randomisation. Older or less fit patients will go directly to a maintenance randomisation.

The value of lenalidomide and lenalidomide combined with vorinostat maintenance will then be assessed by randomising eligible patients to receive either lenalidomide, lenalidomide combined with vorinostat maintenance therapy, or close observation.

The primary end points of the study are overall and progression-free survival (OS and PFS). Secondary end points include response and toxicity.

A number of laboratory based studies will also be performed in order to determine patient specific factors predicting overall and progression-free survival and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or greater
* Newly diagnosed as having symptomatic multiple myeloma or non-secretory multiple myeloma
* Provide written informed consent
* Women of childbearing potential and male patients whose partner is a woman of child bearing potential must be prepared to use contraception in accordance with (and consent to) the Celgene-approved process for thalidomide and lenalidomide Risk Management and Pregnancy Prevention, or commit to absolute and continuous abstinence
* Women of child bearing potential must have a negative pregnancy test performed by a healthcare professional in accordance with the Celgene-approved process for thalidomide and lenalidomide Risk Management and Pregnancy Prevention

Exclusion Criteria:

* Asymptomatic myeloma
* Solitary plasmacytoma of bone. (Patients with previous solitary plasmacytoma now progressed to symptomatic or non-secretory myeloma are eligible)
* Extramedullary plasmacytoma (without evidence of myeloma)
* Previous (<5 years since diagnosis) or concurrent active malignancies, except surgically-removed basal or squamous cell carcinoma of the skin, treated carcinoma in situ of the breast or cervix, or incidental histologic finding of prostate cancer (TMN stage of T1a or 1b). Patients with remote histories (>5 years) of other cured malignancies may be entered.
* Documented diagnosis of Myelodysplastic Syndrome (MDS) that meets International Prognostic Scoring System (IPSS) criteria for high-risk disease
* Previous treatment for myeloma, except the following: local radiotherapy to relieve bone pain or spinal cord compression; or prior bisphosphonate treatment; or corticosteroids within the last 3 months
* Known history of allergy contributable to compounds containing boron or mannitol
* Grade 2 or greater (NCI criteria) peripheral neuropathy
* Acute renal failure (unresponsive to up to 72 hours of rehydration, characterised by creatinine >500µmol/L or urine output <400 mL/day or requirement for dialysis)
* Lactating or breastfeeding
* Patient has active or prior hepatitis C
* Caution is advised in patients with a past history of ischaemic heart disease, pericardial disease, acute diffuse infiltrative pulmonary disease or psychiatric disorders, evidence of impaired marrow function or elevated liver function tests, but exclusion is essentially to be at the discretion of the treating clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4420 (Actual)
Dates: Start 2010-05; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time from initial randomisation to the trial death from any cause or last follow-up
  Overall survival for induction chemotherapy comparisons is defined as the time from initial randomisation to the trial to death from any cause or last follow-up. Overall survival for maintenance therapy comparisons is defined from the time of maintenance randomisation.
Progression-free survival | time from initial randomisation to the trial to progression or death from any cause
  Progression-free survival for induction chemotherapy comparisons is defined as the time from initial randomisation to the trial to progression or death from any cause. Patients who do not progress will be censored at the last date they were known to be alive and progression-free. Progression-free survival for maintenance therapy comparisons is defined from the time of maintenance randomisation

SECONDARY OUTCOMES:
Response | Response will be determined according to the modified international uniform response criteria for multiple myeloma
  Disease progression and response rates will be determined according to the modified International uniform response criteria for multiple myeloma
Toxicity | will be based on adverse events as graded by CTCAE v4.0
  Toxicity will be reported based on adverse events, as graded by CTCAE V4.0 and determined by routine clinical assessments at each centre

CONTACTS AND LOCATIONS:
Overall Officials: Graham Jackson, Principal Investigator — Freeman Health System
Locations (1):
- 112 sites UK wide, United Kingdom, United Kingdom

REFERENCES:
- [Derived] Beer SA, Cairns DA, Pawlyn C, Holroyd A, Ferris E, Cook G, Drayson M, Boyd K, Proszek P, Davies FE, de Tute R, Jenner M, Morgan GJ, Owen R, Hubank M, Houlston R, Jackson G, Kaiser MF. Challenging the concept of functional high-risk myeloma through transcriptional and genetic profiling. Blood. 2025 Nov 27;146(22):2670-2680. doi: 10.1182/blood.2025029987. PMID 40834881
- [Derived] Agbuduwe C, Iqbal G, Cairns D, Menzies T, Dunn J, Gregory W, Kaiser M, Owen R, Pawlyn C, Child JA, Davies F, Morgan GJ, Jackson GH, Drayson MT, Basu S. Clinical characteristics and outcomes of IgD myeloma: experience across UK national trials. Blood Adv. 2022 Sep 13;6(17):5113-5123. doi: 10.1182/bloodadvances.2022007608. PMID 35790108
- [Derived] de Tute RM, Pawlyn C, Cairns DA, Davies FE, Menzies T, Rawstron A, Jones JR, Hockaday A, Henderson R, Cook G, Drayson MT, Jenner MW, Kaiser MF, Gregory WM, Morgan GJ, Jackson GH, Owen RG. Minimal Residual Disease After Autologous Stem-Cell Transplant for Patients With Myeloma: Prognostic Significance and the Impact of Lenalidomide Maintenance and Molecular Risk. J Clin Oncol. 2022 Sep 1;40(25):2889-2900. doi: 10.1200/JCO.21.02228. Epub 2022 Apr 4. PMID 35377708
- [Derived] Walker BA, Boyle EM, Wardell CP, Murison A, Begum DB, Dahir NM, Proszek PZ, Johnson DC, Kaiser MF, Melchor L, Aronson LI, Scales M, Pawlyn C, Mirabella F, Jones JR, Brioli A, Mikulasova A, Cairns DA, Gregory WM, Quartilho A, Drayson MT, Russell N, Cook G, Jackson GH, Leleu X, Davies FE, Morgan GJ. Mutational Spectrum, Copy Number Changes, and Outcome: Results of a Sequencing Study of Patients With Newly Diagnosed Myeloma. J Clin Oncol. 2015 Nov 20;33(33):3911-20. doi: 10.1200/JCO.2014.59.1503. Epub 2015 Aug 17. PMID 26282654
- See also: The ISRCTN register has further information about the Myeloma XI trial. Click on the link above for further information about the trial — http://www.isrctn.com/ISRCTN49407852
- See also: ASCO 2017 abstract: Lenalidomide induction and maintenance therapy for transplant eligible myeloma patients: Results of the Myeloma XI study — http://ascopubs.org/doi/abs/10.1200/JCO.2017.35.15_suppl.8009
- See also: EHA 2017 abstract: QUADRUPLET VS SEQUENTIAL TRIPLET INDUCTION THERAPY FOR MYELOMA PATIENTS: RESULTS OF THE MYELOMA XI STUDY. (EHA-3097) — https://learningcenter.ehaweb.org/eha/2017/22nd/181694/charlotte.pawlyn.quadruplet.vs.sequential.triplet.induction.therapy.for.html
- See also: EHA 2017 abstract: LENALIDOMIDE INDUCTION AND MAINTENANCE THERAPY FOR TRANSPLANT ELIGIBLE MYELOMA: PATIENTS: RESULTS OF THE MYELOMA XI STUDY (EHA-1279) — https://learningcenter.ehaweb.org/eha/2017/22nd/182068/charlotte.pawlyn.lenalidomide.induction.and.maintenance.therapy.for.transplant.html
- See also: Paper in Blood Cancer Journal: Second malignancies in the context of lenalidomide treatment: an analysis of 2732 myeloma patients enrolled to the Myeloma XI trial — http://www.nature.com/articles/bcj2016114